CLINICAL TRIAL: NCT01517789
Title: Advantage of Using Intraoperative Visual Evoked Potentials to Preserve Visual Function During Surgical Procedures Near the Optical Pathways
Acronym: VISUOPEV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHUBX 2011/09
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Surgery; Optic Nerve and Pathway Injury
Keywords: Surgery; Optic Nerve and Pathway Injury; visual event-related potential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental)
  Interventions: Device: Visual evoked potentials monitoring during neurosurgery - Vision monitor MonOpera®

INTERVENTIONS:
Device: Visual evoked potentials monitoring during neurosurgery - Vision monitor MonOpera® — Visual assessment (visual field, visual acuity, pattern visual evoked potential) are realised before and after surgery.
  Flash and steady state visual evoked potential are measured during the surgical procedure at different times.

SUMMARY:
Visual morbidity (visual acuity and/or visual field deficit) must be taken into account during neurosurgical procedures for lesions near the optical pathways. Part of this morbidity is due to surgical manipulation. There is no validated tool for intraoperative visual monitoring and few publications have studied this issue.

In a preliminary work based on analysis of these publications, we defined technical, anaesthetic and analytical parameters in order to optimise intraoperative visual evoked potentials monitoring. These parameters are special devices used for transpalpebral stimulation, complete intravenous anaesthesia without halogen or nitrous oxide, and pertinent analysis criteria of visual evoked potential (VEP). We suppose that these improvements will increase reliability of intraoperative VEP.

DETAILED DESCRIPTION:
This genuine optimised monitoring in France, set up in association with Metrovision company, should help increasing intraoperative VEP reliability as a monitoring tool for visual pathways function.

In this study, we assess the predictive value of relevant intraoperative variations of VEP (more than 50% variation of latency and amplitude) on the visual prognosis at six months after surgery The visual assessment consisting of a visual field, a visual acuity, and the performance of pattern transient VEP, will be performed by an ophthalmologist before surgery, and at three and six months after surgery. An electroencephalogram with photostimulatory lighting will be used in pre-operative and will validate the absence of photo-induced epilepsy risk.

During the intervention, VEPs associated to an electroretinogram will be performed by a neurosurgeon trained to the use of these tools by Metrovision company:

* Under general anaesthesia, but before any surgery.
* During the surgery, at predetermined surgical times (while performing the craniotomy or the sphenoid opening, at various times during the perioptic lesion dissection, after the lesion resection, when closing).

ELIGIBILITY:
Inclusion Criteria:

* Patients with lesion compressing or near the optical pathways

Exclusion Criteria:

* Patients with photic epilepsy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Evolution of visual function six months after surgery. | Month 6 after surgery
  Visual function : visual field and visual acuity six months after surgery.

SECONDARY OUTCOMES:
Score of the visual field. | Month 6 after surgery
Score of visual acuity | Month 6 after surgery
Average diameter of the optic nerve fibers measured with Optical coherence tomography | Month 6 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel LAGUERRE, Dr, Principal Investigator — University Hospital, Bordeaux, France; Paul PEREZ, Dr, Study Chair — University Hospital, Bordeaux, France
Locations (1):
- CHU Bordeaux - hôpital Pellegrin, Bordeaux, France